CLINICAL TRIAL: NCT02414022
Title: Prospective Economic Analysis: A Randomized Phase III CLL Study of Bendamustine Plus Rituximab Versus Ibrutinib + Rituximab vs Ibrutinib Alone in Untreated Older Patients (≥65 Years of Age) With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Economic Analysis of Alliance A041202 CLL Study
Status: Active, not recruiting | Type: Observational
Sponsor: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Other Study IDs: CLC2E
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prospective cost-effectiveness (cost-utility) analysis from the perspective of the Canadian public healthcare system was completed in 2021. Health state utilities were collected using the EuroQOL EQ-5D instrument with Canadian tarrifs applied to calculate quality-adjusted life-years (QALYs). Costs were applied to resource utilization data (expressed in 20196 US dollars). We examined costs and outcomes (QALYs) associated with ibrutinib with rituximab (IR) and BR therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be eligible for the core CLC.2/A041202 protocol.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* Patient must be able (i.e. sufficiently fluent), and willing to complete the health utilities questionnaire in English or French. The baseline assessment must be completed within required timelines, prior to registration/randomization Inability (illiteracy in English or French, loss of sight, or other equivalent reason) to complete the questionnaires will not make the patient ineligible for the core protocol. However, ability but unwillingness to complete the questionnaires will make the patient ineligible for the core protocol.
* Patients must be accessible for treatment and follow-up. Investigators must assure themselves the patients randomized on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.

Exclusion Criteria:

* None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Untreated Older Patients (≥65 Years of Age) with Chronic Lymphocytic Leukemia (CLL)
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2026-04-09 (Estimated)

PRIMARY OUTCOMES:
Measure cost-utility ratio | 5 years
  , as measured in cost per quality-adjusted life-years gained, of ibrutinib-containing regimens compared to bendamustine-rituximab in elderly patients with CLL (Canadian subset of patients). The primary analysis will compare ibrutinib-rituximab with bendamustine-rituximab.

SECONDARY OUTCOMES:
Measure the incremental cost-utility ratio, as measured in cost per quality-adjusted life-years gained, of ibrutinib-alone compared to bendamustine-rituximab in elderly patients with CLL | 5 years
Measure the incremental cost-utility ratio, as measured in cost per quality-adjusted life-years gained, of ibrutinib-rituximab compared to ibrutinib alone in elderly patients with CLL | 5 years
Measure the extended dominance exerted by ibrutinib-rituximab or ibrutinib when compared to bendamustine-rituximab in elderly patients with CLL | 5 years
Measure the incremental cost-effectiveness, as measured in cost per life-years gained, of ibrutinib-containing regimens compared to bendamustine-rituximab in elderly patients with CLL | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Cheung, Study Chair — Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto ON Canada
Locations (15):
- Canada (15):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - The Moncton Hospital, Moncton, New Brunswick
  - Health Sciences North, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Odette Cancer Centre Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network Princess Margaret Cancer Centre, Toronto, Ontario
  - CSSS Champlain-Charles LeMoyne, Greenfield Park, Quebec
  - CHUM-CEntre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Jewish General Hospital, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cheung MC, Mittmann N, Owen C, Abdel-Samad N, Fraser GAM, Lam S, Crump M, Sperlich C, van der Jagt R, Prica A, Couban S, Woyach JA, Ruppert AS, Booth AM, Mandrekar SJ, McDonald G, Shepherd LE, Yen H, Chen BE, Hay AE. A Prospective Economic Analysis of Early Outcome Data From the Alliance A041202/ CCTG CLC.2 Randomized Phase III Trial Of Bendamustine-Rituximab Compared With Ibrutinib-Based Regimens in Untreated Older Patients With Chronic Lymphocytic Leukemia. Clin Lymphoma Myeloma Leuk. 2021 Nov;21(11):766-774. doi: 10.1016/j.clml.2021.06.011. Epub 2021 Jul 3. PMID 34334330